CLINICAL TRIAL: NCT01233648
Title: Resync-AF (Rate vs Rhythm Control in AF Patients With CRT-D)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0601113
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2016-01

CONDITIONS: Atrial Fibrillation
Keywords: heart failure; CRT-D
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Electricity

ARMS (2):
- AF (Active Comparator)
  Interventions: Other: rate control via CRT-D and AVN ablation
- SR (Active Comparator)
  Interventions: Other: rhythm control via pharmacologic, electrical or ablative therapies

INTERVENTIONS:
Other: rate control via CRT-D and AVN ablation — rate control
  Arms: AF
Other: rhythm control via pharmacologic, electrical or ablative therapies — rhythm control
  Arms: SR

SUMMARY:
This study is being done to find out if controlling rate or controlling rhythm is better for heart failure patients who also have AF. Patients with AF who are receiving a CRT-D device and AV node ablation as part of their clinical care will be followed for one year. One group will have their heart rate controlled by the ICD and AVN ablation alone and the second group will be treated with the ICD, AVN ablation and standard medical therapies to restore the heart's normal rhythm. The study doctors will compare the information collected from all of the subjects in this study to see if treating rate or treating rhythm is better in patients with heart failure and AF, resulting in a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Having persistent AF, defined as AF that does not self terminate for at least 24 consecutive hours.
* In AF upon entry into the operating room for CRT-D implantation and AV node ablation.
* Being on a stable dosage of an ACE inhibitor or ARB for at least 1 month preceding implant
* Being on a Beta-blocker for at least 3 months preceding implant and a stable dosage within 1 month of implant
* Not taking or able to be taken off all type I/III antiarrhythmic medications.
* Taking Coumadin so as to maintain an INR of between 2 and 3.
* A Class I or IIa ICD indication
* NYHA Class III/IV within 1 month of baseline
* Intrinsic QRS duration ≥ 130 ms within 1 month prior to baseline
* Left ventricular ejection fraction ≤ 35% (method per physician discretion) within 1 month prior to baseline
* Left ventricular end diastolic dimension (LVEDD) ≥ 55 mm (method per physician discretion) within 1 months prior to baseline
* Willing to provide written informed consent
* Are expected to survive for 6 month of study participation
* Able to tolerate an urgent thoracotomy
* Able to tolerate < 1 mg dexamethasone sodium phosphate (steroid)

Exclusion Criteria:

* Having self-terminating or interminable AF
* Having unstable angina, or having experienced an acute myocardial infarction (MI) or received coronary artery revascularization (CABG) or coronary angioplasty (PTCA) within the past 1 month
* Post-heart transplant (patients on heart transplant list for the first time are not excluded)
* Having mechanical right heart valve
* Having an existing CRT or atrial therapy device(s)
* Being enrolled in any concurrent drug and/or device study which would confound the results of this trial
* Having primary valvular disease and indicated for valve repair or replacement
* Having a previous AV node ablation
* Being on a Type I or Type III anti-arrhythmic medication for the treatment of ventricular tachyarrhythmias
* Women who are pregnant or with child bearing potential and who are not on a reliable form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
AF burden | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David S. Schwartzman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Cardiovascular Institute, Pittsburgh, Pennsylvania, United States